CLINICAL TRIAL: NCT04438005
Title: A Multicenter, Open-Label Study to Investigate the Safety and Efficacy of ICP-022 in Patients With Relapsed/Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: A Study of ICP-022 in Patients With R/R DLBCL
Acronym: DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00108
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Relapsed/Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-022 (Experimental)
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — ICP-022 is a white, round, uncoated tablet, 50 mg. It is administered orally at the dose of 150 mg/day from day 1 to day 28 of each cycle for up to a total of 6 cycles or until progression.

SUMMARY:
It is a phase II, multicenter, open-label study is to evaluate the safety, efficacy and pharmacokinetics of a novel BTK inhibitor, ICP-022, in approximately 85 subjects with R/R DLBCL. There will be no control group in this study. Each subject will receive treatment orally every day in 28-day cycles. Each cycle starts immediately after the previously completed cycle without a break between cycles.

ELIGIBILITY:
Key Inclusion criteria：

1. Men and women between 18 and 75 years old,
2. Histologically confirmed diffuse large B-cell lymphoma（DLBCL）with MyD88 L265P and CD79B positive, at least one measurable tumor of greater than 1.5 centimeter in long axis by contrast-enhanced CT/MRI,
3. ECOG performance status of 0-2,
4. Voluntary written informed consent prior to trail screening.

Key Exclusion criteria:

1. History of other active malignancies, unless cured without evidence of relapse or metastasis within 5 years of study entry
2. History of Richter's syndrome
3. Current or history of lymphoma involved central nervous system
4. Prior corticosteroids (at dosages equivalent to prednisone > 20 mg/day) given with anti-neoplastic intent within 7 days, prior chemotherapy, targeted therapy, radiation therapy, or antibody based therapies or anti-cancer TCM within 4 weeks of the start of study drug.
5. The investigator considers other conditions unsuitable for this study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Overall response rate（ORR） | Up to 3 years
  The efficacy measured by overall response rate (ORR) according to the 2014 International Working Group NHL

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events | Up to 3 years
  The safety of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 5.0 grading criteria
Progression free survival（PFS） | Up to 3 years
  The efficacy measured by progression free survival（PFS）
Duration of response（DOR） | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Affiliated Tumor Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Fourth Hospital of Hebei Medical University, Hebei, Shijiazhuang
  - Hematology Hospital of Chinese Academy of Medical Sciences (Institute of Hematology, Chinese Academy of Medical Sciences), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No